CLINICAL TRIAL: NCT03424785
Title: Long Term Follow-up and Clinical Implications in Chinese Patients With Aortic Intramural Hematoma
Brief Title: Long Term Clinical Implications in Chinese Patients With Aortic Intramural Hematoma
Status: Completed | Type: Observational
Sponsor: Shenyang Northern Hospital (Other)
Responsible Party: Principal Investigator, Han Yaling, MD, Long term follow-up and clinical implications in Chinese patients with aortic intramural hematoma, Shenyang Northern Hospital
Other Study IDs: SYNH-20171115
Record Dates: First submitted 2017-12-11; First posted 2018-02-07 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2017-12

CONDITIONS: Aortic Intramural Hematoma
Keywords: Aortic intramural hematoma; Chinese patients; Clinical outcomes
MeSH Terms: conditions — Aortic Intramural Hematoma | interventions — Pharmaceutical Preparations; Stents; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Imaging Samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: drug, stent, surgical treatment — drug, stent, surgical treatment

SUMMARY:
The study evaluates outcomes of intramural hematomas after long-term follow up and establish predictive factors in Chinese population.

DETAILED DESCRIPTION:
270 intramural hematoma patients with clinical and imaging follow up were retrospectively studied in present study. The primary endpoint was consisted of aortic disease-related death, aortic dissection, penetrating atherosclerotic aortic ulcer , thickening of aorta hematoma and aortic complications requiring surgical or endovascular treatment.

ELIGIBILITY:
Inclusion Criteria:

* Type A aortic hematoma
* Type B aortic hematoma

Exclusion Criteria:

* Aortic without initial intimal flap formation.

Ages: 30 Years to 87 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From February 2003 to May 2017, 1770 consecutive patients were diagnosed with AAS at the General Hospital of Shenyang Military Region, including 270 IMH patients, of which 123 patients were retrospectively examined. Thirty-nine patients presented with type A aortic IMH, and 84 presented with type B aortic IMH
Sampling Method: Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2008-06-03 (Actual); Primary Completion 2017-05-14 (Actual); Study Completion 2017-05-14 (Actual)

PRIMARY OUTCOMES:
hematoma thickness and a baseline MAD | 14years
  Medication and short-term imaging are recommended for Chinese IMH patients with a hematoma thickness less than 10.45 mm and a baseline MAD less than 44.75 mm. Rigorous medical observation should also be performed during the acute phase of IMH.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Harris KM, Braverman AC, Eagle KA, Woznicki EM, Pyeritz RE, Myrmel T, Peterson MD, Voehringer M, Fattori R, Januzzi JL, Gilon D, Montgomery DG, Nienaber CA, Trimarchi S, Isselbacher EM, Evangelista A. Acute aortic intramural hematoma: an analysis from the International Registry of Acute Aortic Dissection. Circulation. 2012 Sep 11;126(11 Suppl 1):S91-6. doi: 10.1161/CIRCULATIONAHA.111.084541. PMID 22965999